Study title: Quantitative Ultrasound with Velacur for Evaluation of Non-Alcoholic Fatty Liver Disease

PI: Samer Gawrieh MD

NCT 04576923

**Statistical Considerations** 

Document date: July 8, 2021

## **Statistical Considerations**

Descriptive statistics such as mean, standard error, and percentages were used to characterize the cohort. Comparisons will be made between groups by using Student t test or analysis of variance. Pearson correlation coefficient will be used to detect the correlation between continuous variables. Multivariate analysis will be performed to examine the independent association between dependent and several independent variables. Sample size is based on clinical experience and precedent established for studies of similar design.